CLINICAL TRIAL: NCT06510400
Title: Clinical Evaluation of Color Stability of Direct Composite Resin Veneers in Vital Anterior Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Abd El Ghany Mohammed, Assistant lecturer, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Color Stability
Record Dates: First submitted 2024-07-14; First posted 2024-07-19 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Tooth Discoloration
MeSH Terms: conditions — Tooth Discoloration

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OMNICHROMA (Experimental): single shade composite was placed to prepared tooth enamel via U veneer template technique
  Interventions: Other: OMNICHROMA; Other: Ceram. x spectra
- Ceram. x spectra (Experimental): multi shade composite was placed to prepared tooth enamel via U veneer template technique
  Interventions: Other: OMNICHROMA; Other: Ceram. x spectra

INTERVENTIONS:
Other: OMNICHROMA — supra nano filled composite
Other: Ceram. x spectra — nano hybrid composite resin

SUMMARY:
Assess color stability of direct veneers over an 18-month recall periods

DETAILED DESCRIPTION:
In today's restorative dentistry, aesthetics has become essential. The primary determinants of the aesthetics of natural teeth are color and form. The significance of color in dental science has greatly increased during the past few decades.

Techniques to restore teeth to their natural appearance have been developed in direct response to patient demand for cosmetic dental procedures. In contemporary cosmetic dentistry, discolorations are often seen as an aesthetic concern.

In order to correct cosmetic flaws in color and form, direct laminate veneers entail the creative application of resin composite material to the tooth surfaces. Because they may be completed chairside, are readily repaired, and have abrasion rates that are similar to those of real teeth, they are viewed as competitors to ceramic veneers.

With direct resin composite veneers, color stability is thought to be a common clinical issue that reduces the aesthetic result over an extended period of clinical service. The capacity of any dental material to retain its original color is known as color stability.

The clinical restoration process is streamlined with the introduction of universal composites, which also considerably reduce chair-side time and simplify the color matching such as OMNICHROMA.

ELIGIBILITY:
Inclusion Criteria:

* have good hygiene.
* No medical diseases
* discolored vital anterior teeth

Exclusion Criteria:

* para functional activities.
* non vital teeth.
* severe intrinsic discoloration.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-07-19 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-04-09 (Actual)

PRIMARY OUTCOMES:
Color stability evaluation | 18 months
  Two calibrated evaluators who were not engaged in the insertion of veneer restorations used VITA Easyshade V to measure the color (ΔE). The device was calibrated before reading.

CONTACTS AND LOCATIONS:
Locations (1):
- Restorative Department, Faculty of Dentistry, Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hirata R, Hilgert LA, Sampaio CS, de Andrade OS, Melo G, Ritter AV. Quo vadis, esthetic dentistry? Part II: Composite resin overtreatment and social media appeal. J Esthet Restor Dent. 2024 Jan;36(1):32-36. doi: 10.1111/jerd.13162. Epub 2023 Dec 23. PMID 38142060
- [Background] de Abreu JLB, Sampaio CS, Benalcazar Jalkh EB, Hirata R. Analysis of the color matching of universal resin composites in anterior restorations. J Esthet Restor Dent. 2021 Mar;33(2):269-276. doi: 10.1111/jerd.12659. Epub 2020 Sep 29. PMID 32989879
- [Background] Fahl N Jr,, Ritter AV. Composite veneers: The direct-indirect technique revisited. J Esthet Restor Dent. 2021 Jan;33(1):7-19. doi: 10.1111/jerd.12696. Epub 2020 Dec 18. PMID 33336852
- [Background] Kam Hepdeniz O, Temel UB. Clinical survival of No-prep indirect composite laminate veneers: a 7-year prospective case series study. BMC Oral Health. 2023 May 3;23(1):257. doi: 10.1186/s12903-023-02949-5. PMID 37138297
- [Background] Zhao X, Zanetti F, Wang L, Pan J, Majeed S, Malmstrom H, Peitsch MC, Hoeng J, Ren Y. Effects of different discoloration challenges and whitening treatments on dental hard tissues and composite resin restorations. J Dent. 2019 Oct;89:103182. doi: 10.1016/j.jdent.2019.103182. Epub 2019 Aug 17. PMID 31430508
- [Background] Miranda AO, Favoreto MW, Matos TP, Castro AS, Kunz P, Souza JL, Carvalho P, Reis A, Loguercio AD. Color Match of a Universal-shade Composite Resin for Restoration of Non-carious Cervical Lesions: An Equivalence Randomized Clinical Trial. Oper Dent. 2024 Jan 1;49(1):20-33. doi: 10.2341/23-021-C. PMID 38057996
- [Background] Huang M, Wang Y, Sun Y, Zhou Y, Liu Y, Ye H. The accuracies of three intraoral scanners with regard to shade determination: An in vitro study. J Prosthodont. 2023 Jun;32(5):111-117. doi: 10.1111/jopr.13571. Epub 2022 Aug 10. PMID 35848886
- [Background] Sabatini C. Color Stability Behavior of Methacrylate-based Resin Composites Polymerized with Light-emitting Diodes and Quartz-Tungsten-Halogen. Oper Dent. 2015 May-Jun;40(3):271-81. doi: 10.2341/14-080-L. Epub 2014 Oct 2. PMID 25275958
- [Background] El-Rashidy AA, Abdelraouf RM, Habib NA. Effect of two artificial aging protocols on color and gloss of single-shade versus multi-shade resin composites. BMC Oral Health. 2022 Aug 1;22(1):321. doi: 10.1186/s12903-022-02351-7. PMID 35915423
- [Background] Mahrous AI, Salama AA, Shabaan AA, Abdou A, Radwan MM. Color stability of two different resin matrix ceramics: randomized clinical trial. BMC Oral Health. 2023 Sep 14;23(1):665. doi: 10.1186/s12903-023-03364-6. PMID 37710194